CLINICAL TRIAL: NCT02636452
Title: Cardiopulmonary Exercise Testing in Interstitial Lung Disease
Status: Completed | Type: Observational
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: 80/2013
Record Dates: First submitted 2015-11-09; First posted 2015-12-21 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: cardiopulmonary exercise test

SUMMARY:
In patients with Interstitial lung diseases (ILD) dyspnea is the most often symptom. Pulmonary lung function tests often do not Show the dyspnea. Aim of the study is to evaluate cardiopulmonary exercise testing concerning therapeutic Monitoring in ILD.

ELIGIBILITY:
Inclusion Criteria:

* informed consent provided
* ILD

Exclusion Criteria:

* no informed consent
* no ILD

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Interstitial lung diseases
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2013-10-31 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Alveolar-arterial oxygen partial pressure difference (AaDO2) in cardipulmonary exercise testing in ILD | quarterly, three years

CONTACTS AND LOCATIONS:
Locations (1):
- Bethanien Hospital, Clinic for Pneumology and Allergology, Center for Sleep and Respiratory Medicine, Solingen, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Fischer A, West SG, Swigris JJ, Brown KK, du Bois RM. Connective tissue disease-associated interstitial lung disease: a call for clarification. Chest. 2010 Aug;138(2):251-6. doi: 10.1378/chest.10-0194. PMID 20682528
- [Result] Fell CD, Liu LX, Motika C, Kazerooni EA, Gross BH, Travis WD, Colby TV, Murray S, Toews GB, Martinez FJ, Flaherty KR. The prognostic value of cardiopulmonary exercise testing in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2009 Mar 1;179(5):402-7. doi: 10.1164/rccm.200802-241OC. Epub 2008 Dec 12. PMID 19074597
- [Derived] Hagmeyer L, Herkenrath S, Anduleit N, Treml M, Randerath W. Cardiopulmonary Exercise Testing Allows Discrimination Between Idiopathic Non-specific Interstitial Pneumonia and Idiopathic Pulmonary Fibrosis in Mild to Moderate Stages of the Disease. Lung. 2019 Dec;197(6):721-726. doi: 10.1007/s00408-019-00282-9. Epub 2019 Nov 1. PMID 31676976